CLINICAL TRIAL: NCT06797661
Title: Insights Into the Pathophysiology of Neurovascular Uncoupling in Patients with Brain Lesions.
Acronym: NVUCVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SRB2024304
Record Dates: First submitted 2025-01-23; First posted 2025-01-28 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma; Glioma; Astrocytoma
Keywords: Primary brain tumor
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma; Brain Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glioma patient (Experimental): As compared to the pre-surgical evaluation that brain tumor patients routinely undergo in our institution, patients are asked to undergo some additional examinations.
  Interventions: Diagnostic Test: Functional MRI; Diagnostic Test: FDG-PET; Diagnostic Test: Structural MRI

INTERVENTIONS:
Diagnostic Test: Functional MRI — 11 minutes of Functional MRI alternating breathing Air-Room and gaz mix (5%CO2 21%O2 74%N2).
  All procedure are acquired simultaneously on a single acquisition on the PET/MRI camera in the institution.
Diagnostic Test: FDG-PET — Some patients who did not benefit from a FDG-PET in their clinical evaluation or more than 1 month before the inclusion in the present study will be ask to also undergo a brain FDG-PET , the dose is set at 2 Mega becquerel per Kg.
  All procedure are acquired simultaneously on a single acquisition on the PET/MRI camera in the institution.
Diagnostic Test: Structural MRI — Patient will benefit Different anatomical sequence of acquisition listed here : T1 , T1 with contrast agent (gadovist) , T2 flair , T2 and DSC (Dynamic susceptibility contrast) , and Time Of Flight .
  All procedure are acquired simultaneously on a single acquisition on the PET/MRI camera in the institution.

SUMMARY:
Neurovascular uncoupling (NVU) represents a major source of potential bias for the identification of eloquent brain regions through activation procedures in blood oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI).

Same region shows proper pattern in glucose metabolism in victiny of brain lesions, investigated with positron emitted tomography with radiolabeled glucose (PET-FDG) This research project aims at investigating the mechanisms of NVU by using a multimodal noninvasive imaging approach in neurosurgical patients.

DETAILED DESCRIPTION:
Brain metabolism and blood flow are tightly coupled with neuronal activity. Changes in neuronal activity result in the modulation of glucose consumption by neurons. Both glucose and lactate levels return to their baseline instantly as neuronal activity ceases, a phenomenon known as neurometabolic coupling. Given the limited energetic reserves in the central nervous system, neuronal activity heavily relies on the finely regulated supply of glucose from the bloodstream. However, the dynamic increase in cerebral blood flow (CBF) during neuronal activation far exceeds the increase in oxidative metabolism. This relative hyperemic response ensures an increased oxygen gradient between blood vessels and tissue, providing ample oxygen supply. The close temporal and regional link between changes in neuronal activity and CBF increase is referred to as neurovascular coupling (NVC) and involves a complex cascade of events. Neurotransmitters, such as glutamate, released at synapses bind to receptors on neurons and astrocytes, leading to the release of various chemical mediators, like nitric oxide and prostaglandins, which directly act on arterial smooth muscle tone. More complex and incompletely understood signaling pathways, including Na+ and Ca2+-mediated astrocyte signaling mechanisms, are also presumed to contribute to NVC.

The tight relationship between neuronal activity and both regional blood flow and metabolism has provided the basis for non-invasive functional brain imaging methods, including positron emission tomography (PET) and functional magnetic resonance imaging (fMRI). PET using [18Fluor ]-fluorodeoxyglucose (FDG) is a technique based on the accumulation of metabolized FDG (i.e., FDG-6-phosphate) in the astrocyte-neuron complex, reflecting the level of glucose consumption. Since the seminal works of Sokoloff et al., glucose utilization is considered a valid, accurate, and quantitative indicator of the level of local neuronal activity within the brain. In contrast, fMRI, which relies on the blood oxygen level-dependent (BOLD) signal, provides indirect information about neuronal activity by investigating perfusion-related changes coupled with neuronal activity. In areas of increased CBF due to modulations in neuronal activity, oxygen delivery exceeds the rate of oxygen utilization, inducing a local increase in the oxy-/deoxy-hemoglobin ratio. This leads to a detectable increase in the magnetic-susceptibility weighted MRI signal.

One of the earliest and still recognized clinical applications of fMRI has been preoperative functional mapping of the primary sensorimotor cortex in patients with brain tumors. This technique has significantly impacted surgical planning, often enabling more aggressive approaches than those considered without functional localization. fMRI has also been increasingly used in the presurgical evaluation of patients with vascular or epileptogenic lesions. However, despite the growing use of BOLD fMRI in patients with brain lesions, this technique has major limitations that must be considered when interpreting fMRI results in such populations. The main limitation is the impairment of BOLD signal changes due to lesion-related loss of normal vascular coupling with neuronal activity, a phenomenon referred to as neurovascular uncoupling (NVU). This can result in false-negative or false-positive results in critical eloquent cortex. If neuronal activity is preserved in diseased but viable cortex, NVU is presumed to occur due to astrocytic, neurotransmitter, or vascular dysfunction.

NVU has been mainly reported in patients with high-grade glial tumors and meningiomas. In such patients, the volume of task-based fMRI signal increases has been shown to be reduced adjacent to the tumor compared to homologous fMRI signal changes in the contralesional hemisphere, despite the absence of neurological deficit. In line with experimental data in healthy subjects showing that BOLD signal may decrease as cerebral blood volume (CBV) increases, impaired cerebrovascular reactivity (CVR) in brain tumor patients may be explained by changes in local perfusion. In hypervascularized tumors such as high-grade gliomas and meningiomas, local hyperperfusion has been suggested to explain the decreased BOLD signal on task-based fMRI. However, recent studies have demonstrated that NVU may also occur in low-grade gliomas. Given the absence of hyperperfusion in this tumor type, different mechanisms need to be considered. In low-grade gliomas, the observed NVU is currently thought to be, at least in part, due to disruption of astrocyte-vascular coupling (gliovascular uncoupling). Patients with arteriovenous malformations may exhibit impaired peri-nidal cerebrovascular reserve due to high-flow shunting, making perfusion-dependent mapping signals unreliable. Epilepsy patients may also exhibit regional impairment of CVR due to dramatic increases in brain metabolism and CBF during the ictal period, disruption of the brain-blood barrier, and an acute loss of cerebral pressure autoregulation.

According to previous research, CVR can be studied through the "hypercapnia challenge" during fMRI recordings, including breath-hold fMRI (BH fMRI) and carbogen inhalation fMRI. Hypercapnia is a potent vasodilator that increases the BOLD baseline signal by detecting an increase in tissue oxygenation resulting from increases in CBF while oxidative metabolism demands are considered to remain constant. However, the influence of hypercapnia on neural activity and neurometabolic/neurovascular couplings is not well understood and remains debated. In practice, areas of reduced or absent hypercapnia-induced increase in fMRI signal on CVR maps compared to homologous contralateral activation are assumed to indicate NVU. Recent studies suggest potential advantages in using resting-state (rs) fMRI as a preoperative technique. rs-fMRI is a functional neuroimaging technique that allows the measurement of spontaneous brain activity in patients at rest. Spontaneous BOLD signal fluctuations are highly correlated in distinct and long-ranged brain regions, indicating functional connectivity within specific and highly organized neuroanatomical networks. Functional connectivity studies have also demonstrated a high degree of spatial correlation between rs-fMRI functional brain connectivity and those studied during a hypercapnia challenge. Interestingly, recent research suggests that rs-BOLD signal may be impaired in patients in whom task-based increases in fMRI signals are reduced or absent due to NVU. Therefore, alterations in functional brain connectivity studied with rs-fMRI might provide insights into the presence of NVU as studied with CVR during hypercapnia. Such findings would be of interest in clinical practice as they could avoid the need for CVR-mapping with a hypercapnia challenge.

ELIGIBILITY:
Inclusion Criteria:

* patients in the study include prior imaging showing a potentially resectable intra-cerebral mass lesion. Patient has to be included before surgery, chemotherapy and radiation

Exclusion Criteria:

* previous brain surgery
* respiratory failure
* Asthma
* Claustrophobia
* Previous adverse reaction to gadovist (contrast agent)
* Pregnancy and Breath feeding
* Diabetes (type I and II)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Effects of Hypercapnia administration on fMRI data | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  For brain fRMI data: BOLD signal variation (Arbitrary Unit from a percent change from baseline).
Effects of Hypercapnia administration on PET-FDG regional standardized data. | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  For brain PET-FDG: regional SUV value (Standardized Uptake Ratio) .The SUV is a mathematically derived ratio of tissue radioactivity concentration at a point in time at a specific region of interest and the injected dose of radioactivity per kilogram of the patient's body weight
Effects of Hypercapnia administration on PET-FDG global data | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  For brain PET-FDG: Statistical Parametric Mapping analysis (SPM) for voxel-wise comparison and multiple correlations (t-score)
Effects of Hypercapnia administration on oxygen saturation (SpO2) | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  SpO2 Variation: Measured in percentage points (%), reflecting the change from baseline levels.
End tidal CO2 | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  End Tidal CO2 during the experiment allow the modelisation and quantification of MRI signal among brain tissue. End tidal CO2 pressure is measured in mmHg
Breathing Rate | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  Breathing Rate during the experiment allow the modelisation and quantification of MRI signal among brain tissue. Breathing rate is measure in respiration per minute
Regional Cerebral Blood Volume | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  CBV represents the volume of blood present in 100 grams of brain tissue at a given time. It is used to assess the vascular capacity of the brain. unit are in mL per 100g of brain tissue .A DSC (Dynamic susceptibility contrast) -MRI is needed, the sequence involves the intravenous injection of a contrast agent, usually gadolinium-based. The contrast agent passes through the brain, and changes in the MRI signal are recorded over time.
Regional Cerebral Blood Flow | end of acquisition ( group of 40 subject estimated at 10 months after first subjet acquisition)
  CBF measures the amount of blood flowing through 100 grams of brain tissue in one minute. This is a crucial measure for assessing cerebral perfusion and identifying areas of under- or hyperperfusion.(mL/100g/min)A DSC-MRI is needed, the sequence involves the intravenous injection of a contrast agent, usually gadolinium-based. The contrast agent passes through the brain, and changes in the MRI signal are recorded over time.

SECONDARY OUTCOMES:
Tumor Grading | up to 2 week after last acquisition to allow Multidisciplinary oncologic commission to fix the grading status
  Tumor Grading, respectively with the World Health Organisation (WHO) 2021 guideline about brain neoplasm
Tumor Histology | up to 2 week after last acquisition to allow Multidisciplinary oncologic commission to fix the grading status
  respectively with the WHO 2021 guideline about brain neoplasm from the surgery clinically planned
Cerebrovascular reactivity mapping | up to 1 month after the last acquisition to allow processing time , all the 40 patient together
  Integration of the variation in fMRI signal and end tidal CO2, and breathing rate into a quantification . The produced data are in % of MRI signal change per mmHg of CO2
Correlation map | up to 1 month after the last acquisition to allow processing time , all the 40 patient together
  Correlation on coregistration of fMRI and PET procedure among the brain and plotted in a linear regression. Correlation will be expressed in Spearman's "R".
Functional connectivity | up to 1 month after the last acquisition to allow processing time , all the 40 patient together
  Measured on resting state data acquired during the experiment , allowing to construct a functional "FC" measure of the hub connected together in the brain. Measured in arbitrary unit.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier De Tiège, MD,PhD, Study Chair — Laboratoire de Neuroanatomie et Neuroimagerie translationnelles Université Libre de Bruxelles
Locations (1):
- HUB-Erasme Hospital, Brussels, Belgium

REFERENCES:
- [Background] Belanger M, Allaman I, Magistretti PJ. Brain energy metabolism: focus on astrocyte-neuron metabolic cooperation. Cell Metab. 2011 Dec 7;14(6):724-38. doi: 10.1016/j.cmet.2011.08.016. PMID 22152301
- [Background] Attwell D, Buchan AM, Charpak S, Lauritzen M, Macvicar BA, Newman EA. Glial and neuronal control of brain blood flow. Nature. 2010 Nov 11;468(7321):232-43. doi: 10.1038/nature09613. PMID 21068832
- [Background] Koehler RC, Roman RJ, Harder DR. Astrocytes and the regulation of cerebral blood flow. Trends Neurosci. 2009 Mar;32(3):160-9. doi: 10.1016/j.tins.2008.11.005. Epub 2009 Jan 21. PMID 19162338
- [Background] Sokoloff L, Reivich M, Kennedy C, Des Rosiers MH, Patlak CS, Pettigrew KD, Sakurada O, Shinohara M. The [14C]deoxyglucose method for the measurement of local cerebral glucose utilization: theory, procedure, and normal values in the conscious and anesthetized albino rat. J Neurochem. 1977 May;28(5):897-916. doi: 10.1111/j.1471-4159.1977.tb10649.x. No abstract available. PMID 864466
- [Background] Ogawa S, Lee TM, Kay AR, Tank DW. Brain magnetic resonance imaging with contrast dependent on blood oxygenation. Proc Natl Acad Sci U S A. 1990 Dec;87(24):9868-72. doi: 10.1073/pnas.87.24.9868. PMID 2124706
- [Background] Sokoloff L. Relation between physiological function and energy metabolism in the central nervous system. J Neurochem. 1977 Jul;29(1):13-26. doi: 10.1111/j.1471-4159.1977.tb03919.x. No abstract available. PMID 407330
- [Background] Buxton RB. The physics of functional magnetic resonance imaging (fMRI). Rep Prog Phys. 2013 Sep;76(9):096601. doi: 10.1088/0034-4885/76/9/096601. Epub 2013 Sep 4. PMID 24006360
- [Background] Mueller WM, Yetkin FZ, Hammeke TA, Morris GL 3rd, Swanson SJ, Reichert K, Cox R, Haughton VM. Functional magnetic resonance imaging mapping of the motor cortex in patients with cerebral tumors. Neurosurgery. 1996 Sep;39(3):515-20; discussion 520-1. doi: 10.1097/00006123-199609000-00015. PMID 8875481
- [Background] Medina LS, Bernal B, Dunoyer C, Cervantes L, Rodriguez M, Pacheco E, Jayakar P, Morrison G, Ragheb J, Altman NR. Seizure disorders: functional MR imaging for diagnostic evaluation and surgical treatment--prospective study. Radiology. 2005 Jul;236(1):247-53. doi: 10.1148/radiol.2361040690. PMID 15987978
- [Background] Petrella JR, Shah LM, Harris KM, Friedman AH, George TM, Sampson JH, Pekala JS, Voyvodic JT. Preoperative functional MR imaging localization of language and motor areas: effect on therapeutic decision making in patients with potentially resectable brain tumors. Radiology. 2006 Sep;240(3):793-802. doi: 10.1148/radiol.2403051153. Epub 2006 Jul 20. PMID 16857981
- [Background] Fierstra J, Conklin J, Krings T, Slessarev M, Han JS, Fisher JA, Terbrugge K, Wallace MC, Tymianski M, Mikulis DJ. Impaired peri-nidal cerebrovascular reserve in seizure patients with brain arteriovenous malformations. Brain. 2011 Jan;134(Pt 1):100-9. doi: 10.1093/brain/awq286. Epub 2010 Nov 24. PMID 21109501
- [Background] Pillai JJ, Williams HT, Faro S. Functional imaging in temporal lobe epilepsy. Semin Ultrasound CT MR. 2007 Dec;28(6):437-50. doi: 10.1053/j.sult.2007.09.006. PMID 18075000
- [Background] Sunaert S. Presurgical planning for tumor resectioning. J Magn Reson Imaging. 2006 Jun;23(6):887-905. doi: 10.1002/jmri.20582. PMID 16649210
- [Background] Holodny AI, Schulder M, Liu WC, Wolko J, Maldjian JA, Kalnin AJ. The effect of brain tumors on BOLD functional MR imaging activation in the adjacent motor cortex: implications for image-guided neurosurgery. AJNR Am J Neuroradiol. 2000 Sep;21(8):1415-22. PMID 11003273
- [Background] Schreiber A, Hubbe U, Ziyeh S, Hennig J. The influence of gliomas and nonglial space-occupying lesions on blood-oxygen-level-dependent contrast enhancement. AJNR Am J Neuroradiol. 2000 Jun-Jul;21(6):1055-63. PMID 10871013
- [Background] Liu WC, Feldman SC, Schulder M, Kalnin AJ, Holodny AI, Zimmerman A, Sinensky R, Rao S. The effect of tumour type and distance on activation in the motor cortex. Neuroradiology. 2005 Nov;47(11):813-9. doi: 10.1007/s00234-005-1428-y. Epub 2005 Sep 2. PMID 16142482
- [Background] Ulmer JL, Hacein-Bey L, Mathews VP, Mueller WM, DeYoe EA, Prost RW, Meyer GA, Krouwer HG, Schmainda KM. Lesion-induced pseudo-dominance at functional magnetic resonance imaging: implications for preoperative assessments. Neurosurgery. 2004 Sep;55(3):569-79; discussion 580-1. doi: 10.1227/01.neu.0000134384.94749.b2. PMID 15335424
- [Background] Fujiwara N, Sakatani K, Katayama Y, Murata Y, Hoshino T, Fukaya C, Yamamoto T. Evoked-cerebral blood oxygenation changes in false-negative activations in BOLD contrast functional MRI of patients with brain tumors. Neuroimage. 2004 Apr;21(4):1464-71. doi: 10.1016/j.neuroimage.2003.10.042. PMID 15050571
- [Background] Krainik A, Duffau H, Capelle L, Cornu P, Boch AL, Mangin JF, Le Bihan D, Marsault C, Chiras J, Lehericy S. Role of the healthy hemisphere in recovery after resection of the supplementary motor area. Neurology. 2004 Apr 27;62(8):1323-32. doi: 10.1212/01.wnl.0000120547.83482.b1. PMID 15111669
- [Background] Hou BL, Bradbury M, Peck KK, Petrovich NM, Gutin PH, Holodny AI. Effect of brain tumor neovasculature defined by rCBV on BOLD fMRI activation volume in the primary motor cortex. Neuroimage. 2006 Aug 15;32(2):489-97. doi: 10.1016/j.neuroimage.2006.04.188. Epub 2006 Jun 27. PMID 16806983
- [Background] Cohen ER, Ugurbil K, Kim SG. Effect of basal conditions on the magnitude and dynamics of the blood oxygenation level-dependent fMRI response. J Cereb Blood Flow Metab. 2002 Sep;22(9):1042-53. doi: 10.1097/00004647-200209000-00002. PMID 12218410
- [Background] Ludemann L, Forschler A, Grieger W, Zimmer C. BOLD signal in the motor cortex shows a correlation with the blood volume of brain tumors. J Magn Reson Imaging. 2006 Apr;23(4):435-43. doi: 10.1002/jmri.20530. PMID 16506145
- [Background] Pillai JJ, Zaca D. Comparison of BOLD cerebrovascular reactivity mapping and DSC MR perfusion imaging for prediction of neurovascular uncoupling potential in brain tumors. Technol Cancer Res Treat. 2012 Aug;11(4):361-74. doi: 10.7785/tcrt.2012.500284. Epub 2012 Mar 1. PMID 22376130
- [Background] Zaca D, Jovicich J, Nadar SR, Voyvodic JT, Pillai JJ. Cerebrovascular reactivity mapping in patients with low grade gliomas undergoing presurgical sensorimotor mapping with BOLD fMRI. J Magn Reson Imaging. 2014 Aug;40(2):383-90. doi: 10.1002/jmri.24406. Epub 2013 Nov 4. PMID 24338845
- [Background] Watkins S, Robel S, Kimbrough IF, Robert SM, Ellis-Davies G, Sontheimer H. Disruption of astrocyte-vascular coupling and the blood-brain barrier by invading glioma cells. Nat Commun. 2014 Jun 19;5:4196. doi: 10.1038/ncomms5196. PMID 24943270
- [Background] Yezhuvath US, Lewis-Amezcua K, Varghese R, Xiao G, Lu H. On the assessment of cerebrovascular reactivity using hypercapnia BOLD MRI. NMR Biomed. 2009 Aug;22(7):779-86. doi: 10.1002/nbm.1392. PMID 19388006
- [Background] Ito H, Kanno I, Ibaraki M, Hatazawa J, Miura S. Changes in human cerebral blood flow and cerebral blood volume during hypercapnia and hypocapnia measured by positron emission tomography. J Cereb Blood Flow Metab. 2003 Jun;23(6):665-70. doi: 10.1097/01.WCB.0000067721.64998.F5. PMID 12796714
- [Background] Hosford PS, Wells JA, Nizari S, Christie IN, Theparambil SM, Castro PA, Hadjihambi A, Barros LF, Ruminot I, Lythgoe MF, Gourine AV. CO2 signaling mediates neurovascular coupling in the cerebral cortex. Nat Commun. 2022 Apr 19;13(1):2125. doi: 10.1038/s41467-022-29622-9. PMID 35440557
- [Background] Zappe AC, Uludag K, Logothetis NK. Direct measurement of oxygen extraction with fMRI using 6% CO2 inhalation. Magn Reson Imaging. 2008 Sep;26(7):961-7. doi: 10.1016/j.mri.2008.02.005. Epub 2008 May 2. PMID 18450401
- [Background] Hall EL, Driver ID, Croal PL, Francis ST, Gowland PA, Morris PG, Brookes MJ. The effect of hypercapnia on resting and stimulus induced MEG signals. Neuroimage. 2011 Oct 15;58(4):1034-43. doi: 10.1016/j.neuroimage.2011.06.073. Epub 2011 Jul 7. PMID 21762783
- [Background] Fox MD, Greicius M. Clinical applications of resting state functional connectivity. Front Syst Neurosci. 2010 Jun 17;4:19. doi: 10.3389/fnsys.2010.00019. eCollection 2010. PMID 20592951
- [Background] Agarwal S, Sair HI, Yahyavi-Firouz-Abadi N, Airan R, Pillai JJ. Neurovascular uncoupling in resting state fMRI demonstrated in patients with primary brain gliomas. J Magn Reson Imaging. 2016 Mar;43(3):620-6. doi: 10.1002/jmri.25012. Epub 2015 Jul 22. PMID 26201672
- [Background] Hou X, Liu P, Gu H, Chan M, Li Y, Peng SL, Wig G, Yang Y, Park D, Lu H. Estimation of brain functional connectivity from hypercapnia BOLD MRI data: Validation in a lifespan cohort of 170 subjects. Neuroimage. 2019 Feb 1;186:455-463. doi: 10.1016/j.neuroimage.2018.11.028. Epub 2018 Nov 18. PMID 30463025
- [Background] Spano VR, Mandell DM, Poublanc J, Sam K, Battisti-Charbonney A, Pucci O, Han JS, Crawley AP, Fisher JA, Mikulis DJ. CO2 blood oxygen level-dependent MR mapping of cerebrovascular reserve in a clinical population: safety, tolerability, and technical feasibility. Radiology. 2013 Feb;266(2):592-8. doi: 10.1148/radiol.12112795. Epub 2012 Nov 30. PMID 23204541